CLINICAL TRIAL: NCT02033434
Title: Pre-hospital Care With Intra-Nasal Ketamine for Transport (PRECINKT): A Pilot Study
Acronym: PRECINKT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. Greg Haljan, Co-principal Investigator, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRECINKT-001
Record Dates: First submitted 2013-12-13; First posted 2014-01-10 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Pain; Traumatic Limb Injury
Keywords: intranasal; ketamine; analgesia; mountain medicine; pre-hospital care; patient transport; pilot study; mountain environment
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intranasal Ketamine (Experimental): All patients
  Interventions: Drug: Intranasal Ketamine

INTERVENTIONS:
Drug: Intranasal Ketamine — Atomized Intranasal Ketamine, 50mg

SUMMARY:
The investigators hypothesize that intra-nasal ketamine, for analgesia of patients with moderate to severe pain in an alpine setting, will provide a clinically significant reduction in pain and provide an effective and feasible alternative to intravenous opioids.

The investigators wish to know:

1. Is our study protocol feasible to study INK in a mountain, prehospital care environment?
2. What estimate can be made of recruitment rates?
3. Does studying the use of INK interfere with or delay care at Whistler/Blackcomb?
4. Is intra-nasal ketamine an effective and safe method for controlling pain in our study population and setting?
5. Does intranasal ketamine provide a clinically significant reduction in pain or do patients require additional IV narcotics for extraction?
6. Are there any significant changes in vital signs after administration of intra-nasal ketamine
7. Does the use of intra-nasal ketamine reduce time of patient extraction and transport in the alpine pre-hospital setting?
8. Are there any long term sequelae of INK at one week?

DETAILED DESCRIPTION:
Whistler/Blackcomb is a large world-class resort that attracts hundreds of thousands of skiers and snowboarders annually for it's steep terrain and excellent on-mountain facilities. Ski patrol operations exist on both mountains and respond to over 10000 injuries per year (1). As both skiing and snowboarding activities gain popularity, the number of people injured also rises (2) as does the demand on ski patrol and attending on-mountain physicians to provide adequate on-mountain treatment.

The provision of analgesia, both to relieve patient suffering and facilitate transport, is a central tenet of pre-hospital care. This is of special import in an alpine setting where environmental factors and challenges with extrication play a significant role in patient outcomes (3). Despite its significance to both patient and practitioner, adequate and timely pain relief is often delayed. The underlying cause is multifactorial; intravenous access is challenging, there is limited availability of advanced health care providers and monitoring capabilities. To date, there remain no widespread guidelines for treatment of acute pain in alpine rescue and ski patrol setting.

Intravenous (IV) opioid analgesia is widely used as a primary method of attaining pain control. While effective, this route of administration has several shortcomings. The insertion of an IV is invasive, painful,, time-consuming, exposes skin to cold injury and delays transport. Opioids also raise the risk of hypotension, hypoxemia and vomiting. In previous work (15), the intranasal (IN) route of medication delivery is rapid, effective and well-tolerated. In addition adverse side effects are minor and transient, and there are no changes in vital signs that required clinical intervention.

This data corroborated previous research that low dose ketamine provides safe and meaningful analgesia while preserving cardiovascular function, respiratory drive and airway reflexes (27). Thus, the use of IN ketamine reduces the need for IV access in stable patients and and reduces the need for monitoring to the risks of opioids (6). These characteristics indicate great potential for ketamine in reducing the extraction and transport time of patients from the mountain environment.

Intranasal ketamine is very attractive in austere and alpine environments, where monitoring capabilities slow transport and IV access is difficult. Previous case reports suggest that IN ketamine provides a rapid, easily administered and effective method of analgesia in the pre-hospital setting (7). However, there is no data on the feasibility of conducting a medical trial in a large busy commercial ski area, nor to calculate an appropriate sample size. The investigators propose a pilot study to investigate the feasibility of conducting a study of IN ketamine (INK) prior to a larger study to determine if INK provides an effective and safe method of analgesia for patients presenting to ski patrol with acute injuries. In addition, although the current body of literature shows minimal adverse events, the investigators will continue to study the safety of INK and monitor for any negative side effects. The purpose is to provide insight and information on the potential utility of IN ketamine in this setting, and to assess feasibility of future clinical trials powered to demonstrate efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* traumatic extremity injury
* age greater than 18 years old
* moderate or severe pain (VNRS 5 or greater)

Exclusion Criteria:

* need for an intravenous catheter as judged by treating physician
* pregnancy
* unable to speak English
* shoulder dislocations,
* previous hypersensitivity, intolerance, or allergy to ketamine,
* structural or functional nasal occlusion,
* inability to understand the VNRS,
* Glasgow Coma Scale <15,
* inability to give informed consent
* history of schizophrenia

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
analgesia | 30 minutes
  clinical effect of intranasal ketamine on pain score measured by verbal analogue scale

SECONDARY OUTCOMES:
transport time | 60 minutes
  the transport time from arrival of first responder to arrival at ambulance pick-up will be compared to historical controls.
cardiorespiratory stability | 30 minutes
  effect of ketamine on heart rate, blood pressure, respiratory rate and oxygen saturation
Satisfaction with medical care and evacuation | 1 week
  Patient, first responder and clinician satisfaction with study protocol and analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Gary Andolfatto, MD, Principal Investigator — University of British Columbia
Locations (1):
- Whistler Blackcomb, Whistler, British Columbia, Canada